CLINICAL TRIAL: NCT01774409
Title: Program to Establish the Genetic and Immunologic Profile of Patient's Tumor for All Types of Advanced Cancer
Acronym: PROFILER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PROFILER; ET12-082 (Other: Sponsor's number)
Record Dates: First submitted 2013-01-16; First posted 2013-01-24 (Estimated); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Neoplasms
Keywords: all advanced malignant tumor
MeSH Terms: conditions — Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Blood and tumor samples (Experimental)
  Interventions: Genetic: Blood and tumor samples

INTERVENTIONS:
Genetic: Blood and tumor samples — Genetic: Establishment of the genetic and immunologic profile
  Whole blood sampling :
  * 1 tube for the constitutional DNA extraction;
  * 3 tubes for ancillary studies and research.
  Collection of the available archival tumor sample (frozen or FFPE). If there's no available sample, the investigator will prescribe a biopsy of a reachable lesion.
  With the established profile, recommendations will be given by a multidisciplinary molecular board.

SUMMARY:
It is a non-randomized, multicentric, cohort study, combined with a biological sample collection, a clinical data collection and with a genetic and immunologic biomarkers study.

The ProfiLER program aims to implement a personalized cancer medicine approach by proposing to establish the genetic and immunologic profile of the tumor for patients with an advanced malignant tumor, in order to define a map of genetic (for the pre-identified target genes) and immunologic profiles for all the studied types of cancer. This study will also allow adapting the therapeutic management of these patients, if needed, by giving them targeted therapies or immunotherapies (commercialized on in ongoing clinical trials), based on the recommendations of the multidisciplinary molecular board.

The genetic and immunologic profile of the tumor will be determined from archival or fresh collected (biopsy of a reachable lesion) tumor sample and from a blood sample. The correlation between genetic profiles of the tumor, patients immunity status and clinical data (progression, tumor response, etc.) collected from the patient medical records will probably allow us to identify biomarkers with a potential predictive value and to determine if some genetic disorders are linked to immunity status alterations.

DETAILED DESCRIPTION:
Determination of the tumor profile and review in multidisciplinary molecular board:

The genetic and immunologic profile will be performed from the available tumor sample and from a blood sample.

Genetic profile:

* Research of mutations/insertions/deletions for an array of predefined genes in tumor deoxyribonucleic acid by high-throughput sequencing
* Analysis of copy number variations of genes on tumor deoxyribonucleic acid by microarray-based comparative genomic hybridization
* Analysis of rearrangements involving the gene Anaplastic Lymphoma Kinase that can't be detected by Next Generation Sequencing or array Comparative Genomic Hybridization (balanced translocations) by means of fluorescent hybridization probes on tumor samples Immunologic profile: analysis of the expression of relevant immunologic markers

Clinical data collection:

Patients' clinical data will be collected from the patient medical record. This study is not a treatment evaluation. Patients' follow-up and treatment will be performed according to the center local practices or to the specificities of a clinical trial in which the patient would have been enrolled, depending on the recommendations given by the multidisciplinary molecular board, with the review of the tumor genetic profile.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of advanced (locally-advanced or metastatic) malignant tumor of any histological type
* Tumor sample available to determine the genetic profile: either archival tumor sample [FFPE (formalin fixed and paraffin embedded)] or perform a new biopsy on an accessible lesion (left at the investigator's appreciation). For biopsies, presence of at least one tumor lesion with a diameter ≥ 20 mm, visible by medical imaging and accessible to repeatable percutaneous (needle biopsies 18 gauge or larger) sampling that permit core needle biopsy (ideally 4 cores) without unacceptable risk of a major procedural complication. Please note that brain and bone lesions are not considered as accessible lesions.
* Patient with 1st, 2nd or 3rd line therapy (NB: endocrine therapy (monotherapy) are not considered as line therapy) for advanced / metastatic cancer.
* For patients over 70 years of age, a Performance Status (PS) of 0 on the ECOG scale.
* Patient must be covered by a medical insurance.
* Informed consent signed by the patient and/or by parents (or legal representative) for patients below 18.

Exclusion Criteria:

* No tumor sample available.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2013-02; Primary Completion 2025-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Establish a map of genetic profiles (for the pre-identified target genes) for all types of advanced malignant tumors. | at least 3 years after patient enrollment
  Description of the incidence rates of each detected genetic disorder among the pre-identified target genes in the global cohort and for each histological type.

SECONDARY OUTCOMES:
Establish a map of immunologic profiles for all types of advanced malignant tumors. | at least 3 years after patient enrollment
  Description of the incidence rates of each detected immunologic disorder in the global cohort and for each histological type.
Determine for each histological type of tumor, characteristic profiles of genetic and/or immunologic disorders and disorders that might be common to several histological types. | at least 3 years after patient enrollment
  Comparison of the genetic and immunologic profiles between patients with the same tumor type or between tumors of different types.
Identify genetic and/or immunologic biomarkers (or molecular profiles) with a potential predictive value on response to treatments. | at least 3 years after patient enrollment
  Tumor response (determined by the investigator and/or the radiologist) assessed after each treatment received by the patient during his/her whole participation to the study (if data are available in the medical record).
Identify biomarkers (constitutional or somatic alterations in tumor cells) that might be correlated with systemic or local alterations of the immunity status observed in some patients with advanced cancers | at least 3 years after patient enrollment
  lymphopenia, over-representation of Treg, dendritic cells alterations,
Assess the changes of genetic and/or immunologic profiles in case of progressive disease | at least 3 years after patient enrollment
Number of patients with a recommanded therapy based on their molecular profil and/or for whom the therapy hs been administrated and description of the recommanded therapy | at least 3 years after patient enrollment
  A description will be done of therapie(s) recommanded and/or received by patients based on recommandation done by the Molecular Tumor Board after reviewing of molecular profil
Describe the clinical impact of this molecular profiling in term of PFS | at least 3 years after patient enrollment
  Progression free survival for each recommanded therapies received
Describe the clinical impact of this molecular profiling in term of OS | at least 3 years after patient enrollment
  Overall survival for each recommanded therapies received
Describe the clinical impact of this molecular profiling in term of tumor response | at least 3 years after patient enrollment
  Tumoral response (clinic and/or radiologic) for each recommanded therapies received

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Yves BLAY, MD PhD, Principal Investigator — Centre Leon Berard
Locations (6):
- France (6):
  - Centre Hospitalier Annecy Genevois, Annecy
  - Groupement Hospitalier Mutualiste, Grenoble
  - Hôpital Edouard Herriot, Lyon
  - Centre Léon Bérard, Lyon
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU de Saint-Etienne Hôpital Nord, Saint-Etienne

REFERENCES:
- [Background] Stratton MR, Campbell PJ, Futreal PA. The cancer genome. Nature. 2009 Apr 9;458(7239):719-24. doi: 10.1038/nature07943. PMID 19360079
- [Background] Diaz-Cano SJ. General morphological and biological features of neoplasms: integration of molecular findings. Histopathology. 2008 Jul;53(1):1-19. doi: 10.1111/j.1365-2559.2007.02937.x. Epub 2008 Feb 12. PMID 18282144
- [Background] Dancey JE, Bedard PL, Onetto N, Hudson TJ. The genetic basis for cancer treatment decisions. Cell. 2012 Feb 3;148(3):409-20. doi: 10.1016/j.cell.2012.01.014. PMID 22304912
- [Background] Chin L, Hahn WC, Getz G, Meyerson M. Making sense of cancer genomic data. Genes Dev. 2011 Mar 15;25(6):534-55. doi: 10.1101/gad.2017311. PMID 21406553
- [Background] International Cancer Genome Consortium; Hudson TJ, Anderson W, Artez A, Barker AD, Bell C, Bernabe RR, Bhan MK, Calvo F, Eerola I, Gerhard DS, Guttmacher A, Guyer M, Hemsley FM, Jennings JL, Kerr D, Klatt P, Kolar P, Kusada J, Lane DP, Laplace F, Youyong L, Nettekoven G, Ozenberger B, Peterson J, Rao TS, Remacle J, Schafer AJ, Shibata T, Stratton MR, Vockley JG, Watanabe K, Yang H, Yuen MM, Knoppers BM, Bobrow M, Cambon-Thomsen A, Dressler LG, Dyke SO, Joly Y, Kato K, Kennedy KL, Nicolas P, Parker MJ, Rial-Sebbag E, Romeo-Casabona CM, Shaw KM, Wallace S, Wiesner GL, Zeps N, Lichter P, Biankin AV, Chabannon C, Chin L, Clement B, de Alava E, Degos F, Ferguson ML, Geary P, Hayes DN, Hudson TJ, Johns AL, Kasprzyk A, Nakagawa H, Penny R, Piris MA, Sarin R, Scarpa A, Shibata T, van de Vijver M, Futreal PA, Aburatani H, Bayes M, Botwell DD, Campbell PJ, Estivill X, Gerhard DS, Grimmond SM, Gut I, Hirst M, Lopez-Otin C, Majumder P, Marra M, McPherson JD, Nakagawa H, Ning Z, Puente XS, Ruan Y, Shibata T, Stratton MR, Stunnenberg HG, Swerdlow H, Velculescu VE, Wilson RK, Xue HH, Yang L, Spellman PT, Bader GD, Boutros PC, Campbell PJ, Flicek P, Getz G, Guigo R, Guo G, Haussler D, Heath S, Hubbard TJ, Jiang T, Jones SM, Li Q, Lopez-Bigas N, Luo R, Muthuswamy L, Ouellette BF, Pearson JV, Puente XS, Quesada V, Raphael BJ, Sander C, Shibata T, Speed TP, Stein LD, Stuart JM, Teague JW, Totoki Y, Tsunoda T, Valencia A, Wheeler DA, Wu H, Zhao S, Zhou G, Stein LD, Guigo R, Hubbard TJ, Joly Y, Jones SM, Kasprzyk A, Lathrop M, Lopez-Bigas N, Ouellette BF, Spellman PT, Teague JW, Thomas G, Valencia A, Yoshida T, Kennedy KL, Axton M, Dyke SO, Futreal PA, Gerhard DS, Gunter C, Guyer M, Hudson TJ, McPherson JD, Miller LJ, Ozenberger B, Shaw KM, Kasprzyk A, Stein LD, Zhang J, Haider SA, Wang J, Yung CK, Cros A, Liang Y, Gnaneshan S, Guberman J, Hsu J, Bobrow M, Chalmers DR, Hasel KW, Joly Y, Kaan TS, Kennedy KL, Knoppers BM, Lowrance WW, Masui T, Nicolas P, Rial-Sebbag E, Rodriguez LL, Vergely C, Yoshida T, Grimmond SM, Biankin AV, Bowtell DD, Cloonan N, deFazio A, Eshleman JR, Etemadmoghadam D, Gardiner BB, Kench JG, Scarpa A, Sutherland RL, Tempero MA, Waddell NJ, Wilson PJ, McPherson JD, Gallinger S, Tsao MS, Shaw PA, Petersen GM, Mukhopadhyay D, Chin L, DePinho RA, Thayer S, Muthuswamy L, Shazand K, Beck T, Sam M, Timms L, Ballin V, Lu Y, Ji J, Zhang X, Chen F, Hu X, Zhou G, Yang Q, Tian G, Zhang L, Xing X, Li X, Zhu Z, Yu Y, Yu J, Yang H, Lathrop M, Tost J, Brennan P, Holcatova I, Zaridze D, Brazma A, Egevard L, Prokhortchouk E, Banks RE, Uhlen M, Cambon-Thomsen A, Viksna J, Ponten F, Skryabin K, Stratton MR, Futreal PA, Birney E, Borg A, Borresen-Dale AL, Caldas C, Foekens JA, Martin S, Reis-Filho JS, Richardson AL, Sotiriou C, Stunnenberg HG, Thoms G, van de Vijver M, van't Veer L, Calvo F, Birnbaum D, Blanche H, Boucher P, Boyault S, Chabannon C, Gut I, Masson-Jacquemier JD, Lathrop M, Pauporte I, Pivot X, Vincent-Salomon A, Tabone E, Theillet C, Thomas G, Tost J, Treilleux I, Calvo F, Bioulac-Sage P, Clement B, Decaens T, Degos F, Franco D, Gut I, Gut M, Heath S, Lathrop M, Samuel D, Thomas G, Zucman-Rossi J, Lichter P, Eils R, Brors B, Korbel JO, Korshunov A, Landgraf P, Lehrach H, Pfister S, Radlwimmer B, Reifenberger G, Taylor MD, von Kalle C, Majumder PP, Sarin R, Rao TS, Bhan MK, Scarpa A, Pederzoli P, Lawlor RA, Delledonne M, Bardelli A, Biankin AV, Grimmond SM, Gress T, Klimstra D, Zamboni G, Shibata T, Nakamura Y, Nakagawa H, Kusada J, Tsunoda T, Miyano S, Aburatani H, Kato K, Fujimoto A, Yoshida T, Campo E, Lopez-Otin C, Estivill X, Guigo R, de Sanjose S, Piris MA, Montserrat E, Gonzalez-Diaz M, Puente XS, Jares P, Valencia A, Himmelbauer H, Quesada V, Bea S, Stratton MR, Futreal PA, Campbell PJ, Vincent-Salomon A, Richardson AL, Reis-Filho JS, van de Vijver M, Thomas G, Masson-Jacquemier JD, Aparicio S, Borg A, Borresen-Dale AL, Caldas C, Foekens JA, Stunnenberg HG, van't Veer L, Easton DF, Spellman PT, Martin S, Barker AD, Chin L, Collins FS, Compton CC, Ferguson ML, Gerhard DS, Getz G, Gunter C, Guttmacher A, Guyer M, Hayes DN, Lander ES, Ozenberger B, Penny R, Peterson J, Sander C, Shaw KM, Speed TP, Spellman PT, Vockley JG, Wheeler DA, Wilson RK, Hudson TJ, Chin L, Knoppers BM, Lander ES, Lichter P, Stein LD, Stratton MR, Anderson W, Barker AD, Bell C, Bobrow M, Burke W, Collins FS, Compton CC, DePinho RA, Easton DF, Futreal PA, Gerhard DS, Green AR, Guyer M, Hamilton SR, Hubbard TJ, Kallioniemi OP, Kennedy KL, Ley TJ, Liu ET, Lu Y, Majumder P, Marra M, Ozenberger B, Peterson J, Schafer AJ, Spellman PT, Stunnenberg HG, Wainwright BJ, Wilson RK, Yang H. International network of cancer genome projects. Nature. 2010 Apr 15;464(7291):993-8. doi: 10.1038/nature08987. PMID 20393554
- [Background] Davies H, Bignell GR, Cox C, Stephens P, Edkins S, Clegg S, Teague J, Woffendin H, Garnett MJ, Bottomley W, Davis N, Dicks E, Ewing R, Floyd Y, Gray K, Hall S, Hawes R, Hughes J, Kosmidou V, Menzies A, Mould C, Parker A, Stevens C, Watt S, Hooper S, Wilson R, Jayatilake H, Gusterson BA, Cooper C, Shipley J, Hargrave D, Pritchard-Jones K, Maitland N, Chenevix-Trench G, Riggins GJ, Bigner DD, Palmieri G, Cossu A, Flanagan A, Nicholson A, Ho JW, Leung SY, Yuen ST, Weber BL, Seigler HF, Darrow TL, Paterson H, Marais R, Marshall CJ, Wooster R, Stratton MR, Futreal PA. Mutations of the BRAF gene in human cancer. Nature. 2002 Jun 27;417(6892):949-54. doi: 10.1038/nature00766. Epub 2002 Jun 9. PMID 12068308
- [Background] Samuels Y, Wang Z, Bardelli A, Silliman N, Ptak J, Szabo S, Yan H, Gazdar A, Powell SM, Riggins GJ, Willson JK, Markowitz S, Kinzler KW, Vogelstein B, Velculescu VE. High frequency of mutations of the PIK3CA gene in human cancers. Science. 2004 Apr 23;304(5670):554. doi: 10.1126/science.1096502. Epub 2004 Mar 11. No abstract available. PMID 15016963
- [Background] Arteaga CL, Baselga J. Impact of genomics on personalized cancer medicine. Clin Cancer Res. 2012 Feb 1;18(3):612-8. doi: 10.1158/1078-0432.CCR-11-2019. PMID 22298893
- [Background] Pao W, Wang TY, Riely GJ, Miller VA, Pan Q, Ladanyi M, Zakowski MF, Heelan RT, Kris MG, Varmus HE. KRAS mutations and primary resistance of lung adenocarcinomas to gefitinib or erlotinib. PLoS Med. 2005 Jan;2(1):e17. doi: 10.1371/journal.pmed.0020017. Epub 2005 Jan 25. PMID 15696205
- [Background] Lievre A, Bachet JB, Le Corre D, Boige V, Landi B, Emile JF, Cote JF, Tomasic G, Penna C, Ducreux M, Rougier P, Penault-Llorca F, Laurent-Puig P. KRAS mutation status is predictive of response to cetuximab therapy in colorectal cancer. Cancer Res. 2006 Apr 15;66(8):3992-5. doi: 10.1158/0008-5472.CAN-06-0191. PMID 16618717
- [Background] Macconaill LE, Garraway LA. Clinical implications of the cancer genome. J Clin Oncol. 2010 Dec 10;28(35):5219-28. doi: 10.1200/JCO.2009.27.4944. Epub 2010 Oct 25. PMID 20975063
- [Background] Ray-Coquard I, Ghesquiere H, Bachelot T, Borg C, Biron P, Sebban C, LeCesne A, Chauvin F, Blay JY; ELYPSE Study Group. Identification of patients at risk for early death after conventional chemotherapy in solid tumours and lymphomas. Br J Cancer. 2001 Sep 14;85(6):816-22. doi: 10.1054/bjoc.2001.2011. PMID 11556830
- [Background] Borg C, Ray-Coquard I, Philip I, Clapisson G, Bendriss-Vermare N, Menetrier-Caux C, Sebban C, Biron P, Blay JY. CD4 lymphopenia as a risk factor for febrile neutropenia and early death after cytotoxic chemotherapy in adult patients with cancer. Cancer. 2004 Dec 1;101(11):2675-80. doi: 10.1002/cncr.20688. PMID 15503313
- [Background] Ray-Coquard I, Cropet C, Van Glabbeke M, Sebban C, Le Cesne A, Judson I, Tredan O, Verweij J, Biron P, Labidi I, Guastalla JP, Bachelot T, Perol D, Chabaud S, Hogendoorn PC, Cassier P, Dufresne A, Blay JY; European Organization for Research and Treatment of Cancer Soft Tissue and Bone Sarcoma Group. Lymphopenia as a prognostic factor for overall survival in advanced carcinomas, sarcomas, and lymphomas. Cancer Res. 2009 Jul 1;69(13):5383-91. doi: 10.1158/0008-5472.CAN-08-3845. Epub 2009 Jun 23. PMID 19549917
- [Background] Manuel M, Tredan O, Bachelot T, Clapisson G, Courtier A, Parmentier G, Rabeony T, Grives A, Perez S, Mouret JF, Perol D, Chabaud S, Ray-Coquard I, Labidi-Galy I, Heudel P, Pierga JY, Caux C, Blay JY, Pasqual N, Menetrier-Caux C. Lymphopenia combined with low TCR diversity (divpenia) predicts poor overall survival in metastatic breast cancer patients. Oncoimmunology. 2012 Jul 1;1(4):432-440. doi: 10.4161/onci.19545. PMID 22754761
- [Background] Menetrier-Caux C, Gobert M, Caux C. Differences in tumor regulatory T-cell localization and activation status impact patient outcome. Cancer Res. 2009 Oct 15;69(20):7895-8. doi: 10.1158/0008-5472.CAN-09-1642. Epub 2009 Oct 6. PMID 19808962
- [Background] Labidi-Galy SI, Sisirak V, Meeus P, Gobert M, Treilleux I, Bajard A, Combes JD, Faget J, Mithieux F, Cassignol A, Tredan O, Durand I, Menetrier-Caux C, Caux C, Blay JY, Ray-Coquard I, Bendriss-Vermare N. Quantitative and functional alterations of plasmacytoid dendritic cells contribute to immune tolerance in ovarian cancer. Cancer Res. 2011 Aug 15;71(16):5423-34. doi: 10.1158/0008-5472.CAN-11-0367. Epub 2011 Jun 22. PMID 21697280
- [Background] Sisirak V, Faget J, Gobert M, Goutagny N, Vey N, Treilleux I, Renaudineau S, Poyet G, Labidi-Galy SI, Goddard-Leon S, Durand I, Le Mercier I, Bajard A, Bachelot T, Puisieux A, Puisieux I, Blay JY, Menetrier-Caux C, Caux C, Bendriss-Vermare N. Impaired IFN-alpha production by plasmacytoid dendritic cells favors regulatory T-cell expansion that may contribute to breast cancer progression. Cancer Res. 2012 Oct 15;72(20):5188-97. doi: 10.1158/0008-5472.CAN-11-3468. Epub 2012 Jul 25. PMID 22836755
- [Background] Thompson RH, Gillett MD, Cheville JC, Lohse CM, Dong H, Webster WS, Krejci KG, Lobo JR, Sengupta S, Chen L, Zincke H, Blute ML, Strome SE, Leibovich BC, Kwon ED. Costimulatory B7-H1 in renal cell carcinoma patients: Indicator of tumor aggressiveness and potential therapeutic target. Proc Natl Acad Sci U S A. 2004 Dec 7;101(49):17174-9. doi: 10.1073/pnas.0406351101. Epub 2004 Nov 29. PMID 15569934
- [Background] Hamanishi J, Mandai M, Iwasaki M, Okazaki T, Tanaka Y, Yamaguchi K, Higuchi T, Yagi H, Takakura K, Minato N, Honjo T, Fujii S. Programmed cell death 1 ligand 1 and tumor-infiltrating CD8+ T lymphocytes are prognostic factors of human ovarian cancer. Proc Natl Acad Sci U S A. 2007 Feb 27;104(9):3360-5. doi: 10.1073/pnas.0611533104. Epub 2007 Feb 21. PMID 17360651
- [Background] Brahmer JR, Tykodi SS, Chow LQ, Hwu WJ, Topalian SL, Hwu P, Drake CG, Camacho LH, Kauh J, Odunsi K, Pitot HC, Hamid O, Bhatia S, Martins R, Eaton K, Chen S, Salay TM, Alaparthy S, Grosso JF, Korman AJ, Parker SM, Agrawal S, Goldberg SM, Pardoll DM, Gupta A, Wigginton JM. Safety and activity of anti-PD-L1 antibody in patients with advanced cancer. N Engl J Med. 2012 Jun 28;366(26):2455-65. doi: 10.1056/NEJMoa1200694. Epub 2012 Jun 2. PMID 22658128
- [Background] Topalian SL, Hodi FS, Brahmer JR, Gettinger SN, Smith DC, McDermott DF, Powderly JD, Carvajal RD, Sosman JA, Atkins MB, Leming PD, Spigel DR, Antonia SJ, Horn L, Drake CG, Pardoll DM, Chen L, Sharfman WH, Anders RA, Taube JM, McMiller TL, Xu H, Korman AJ, Jure-Kunkel M, Agrawal S, McDonald D, Kollia GD, Gupta A, Wigginton JM, Sznol M. Safety, activity, and immune correlates of anti-PD-1 antibody in cancer. N Engl J Med. 2012 Jun 28;366(26):2443-54. doi: 10.1056/NEJMoa1200690. Epub 2012 Jun 2. PMID 22658127
- [Background] Pavlidis N, Hansen H, Stahel R. ESMO Clinical Practice Guidelines: development, implementation and dissemination. Ann Oncol. 2010 May;21 Suppl 5:v7-8. doi: 10.1093/annonc/mdq158. No abstract available. PMID 20555106
- [Background] Kantarjian H, Sawyers C, Hochhaus A, Guilhot F, Schiffer C, Gambacorti-Passerini C, Niederwieser D, Resta D, Capdeville R, Zoellner U, Talpaz M, Druker B, Goldman J, O'Brien SG, Russell N, Fischer T, Ottmann O, Cony-Makhoul P, Facon T, Stone R, Miller C, Tallman M, Brown R, Schuster M, Loughran T, Gratwohl A, Mandelli F, Saglio G, Lazzarino M, Russo D, Baccarani M, Morra E; International STI571 CML Study Group. Hematologic and cytogenetic responses to imatinib mesylate in chronic myelogenous leukemia. N Engl J Med. 2002 Feb 28;346(9):645-52. doi: 10.1056/NEJMoa011573. PMID 11870241
- [Background] Demetri GD, von Mehren M, Blanke CD, Van den Abbeele AD, Eisenberg B, Roberts PJ, Heinrich MC, Tuveson DA, Singer S, Janicek M, Fletcher JA, Silverman SG, Silberman SL, Capdeville R, Kiese B, Peng B, Dimitrijevic S, Druker BJ, Corless C, Fletcher CD, Joensuu H. Efficacy and safety of imatinib mesylate in advanced gastrointestinal stromal tumors. N Engl J Med. 2002 Aug 15;347(7):472-80. doi: 10.1056/NEJMoa020461. PMID 12181401
- [Background] Heinrich MC, Corless CL, Demetri GD, Blanke CD, von Mehren M, Joensuu H, McGreevey LS, Chen CJ, Van den Abbeele AD, Druker BJ, Kiese B, Eisenberg B, Roberts PJ, Singer S, Fletcher CD, Silberman S, Dimitrijevic S, Fletcher JA. Kinase mutations and imatinib response in patients with metastatic gastrointestinal stromal tumor. J Clin Oncol. 2003 Dec 1;21(23):4342-9. doi: 10.1200/JCO.2003.04.190. PMID 14645423
- [Background] Debiec-Rychter M, Sciot R, Le Cesne A, Schlemmer M, Hohenberger P, van Oosterom AT, Blay JY, Leyvraz S, Stul M, Casali PG, Zalcberg J, Verweij J, Van Glabbeke M, Hagemeijer A, Judson I; EORTC Soft Tissue and Bone Sarcoma Group; Italian Sarcoma Group; Australasian GastroIntestinal Trials Group. KIT mutations and dose selection for imatinib in patients with advanced gastrointestinal stromal tumours. Eur J Cancer. 2006 May;42(8):1093-103. doi: 10.1016/j.ejca.2006.01.030. Epub 2006 Apr 18. PMID 16624552
- [Background] Guo J, Si L, Kong Y, Flaherty KT, Xu X, Zhu Y, Corless CL, Li L, Li H, Sheng X, Cui C, Chi Z, Li S, Han M, Mao L, Lin X, Du N, Zhang X, Li J, Wang B, Qin S. Phase II, open-label, single-arm trial of imatinib mesylate in patients with metastatic melanoma harboring c-Kit mutation or amplification. J Clin Oncol. 2011 Jul 20;29(21):2904-9. doi: 10.1200/JCO.2010.33.9275. Epub 2011 Jun 20. PMID 21690468
- [Background] Dienstmann R, Tabernero J. BRAF as a target for cancer therapy. Anticancer Agents Med Chem. 2011 Mar;11(3):285-95. doi: 10.2174/187152011795347469. PMID 21426297
- [Background] Chapman PB, Hauschild A, Robert C, Haanen JB, Ascierto P, Larkin J, Dummer R, Garbe C, Testori A, Maio M, Hogg D, Lorigan P, Lebbe C, Jouary T, Schadendorf D, Ribas A, O'Day SJ, Sosman JA, Kirkwood JM, Eggermont AM, Dreno B, Nolop K, Li J, Nelson B, Hou J, Lee RJ, Flaherty KT, McArthur GA; BRIM-3 Study Group. Improved survival with vemurafenib in melanoma with BRAF V600E mutation. N Engl J Med. 2011 Jun 30;364(26):2507-16. doi: 10.1056/NEJMoa1103782. Epub 2011 Jun 5. PMID 21639808
- [Background] Kwak EL, Bang YJ, Camidge DR, Shaw AT, Solomon B, Maki RG, Ou SH, Dezube BJ, Janne PA, Costa DB, Varella-Garcia M, Kim WH, Lynch TJ, Fidias P, Stubbs H, Engelman JA, Sequist LV, Tan W, Gandhi L, Mino-Kenudson M, Wei GC, Shreeve SM, Ratain MJ, Settleman J, Christensen JG, Haber DA, Wilner K, Salgia R, Shapiro GI, Clark JW, Iafrate AJ. Anaplastic lymphoma kinase inhibition in non-small-cell lung cancer. N Engl J Med. 2010 Oct 28;363(18):1693-703. doi: 10.1056/NEJMoa1006448. PMID 20979469
- [Background] Arteaga CL, Sliwkowski MX, Osborne CK, Perez EA, Puglisi F, Gianni L. Treatment of HER2-positive breast cancer: current status and future perspectives. Nat Rev Clin Oncol. 2011 Nov 29;9(1):16-32. doi: 10.1038/nrclinonc.2011.177. PMID 22124364
- [Derived] Benezech S, Saintigny P, Attignon V, Pissaloux D, Paindavoine S, Faure-Conter C, Corradini N, Marec-Berard P, Bergeron C, Cassier P, Eberst L, Dufresne A, Wang Q, Agrapart V, De La Fouchardiere A, Perol D, Garin G, Corset V, Ben Abdesselem L, Chabaud S, Tredan O, Blay JY, Frappaz D. Tumor Molecular Profiling: Pediatric Results of the ProfiLER Study. JCO Precis Oncol. 2020 Nov;4:785-795. doi: 10.1200/PO.20.00023. PMID 35050753
- [Derived] Tredan O, Wang Q, Pissaloux D, Cassier P, de la Fouchardiere A, Fayette J, Desseigne F, Ray-Coquard I, de la Fouchardiere C, Frappaz D, Heudel PE, Bonneville-Levard A, Flechon A, Sarabi M, Guibert P, Bachelot T, Perol M, You B, Bonnin N, Collard O, Leyronnas C, Attignon V, Baudet C, Sohier E, Villemin JP, Viari A, Boyault S, Lantuejoul S, Paindavoine S, Treillleux I, Rodriguez C, Agrapart V, Corset V, Garin G, Chabaud S, Perol D, Blay JY; ProfiLER investigators. Molecular screening program to select molecular-based recommended therapies for metastatic cancer patients: analysis from the ProfiLER trial. Ann Oncol. 2019 May 1;30(5):757-765. doi: 10.1093/annonc/mdz080. PMID 30865223
- [Derived] Jiang X, Pissaloux D, De La Fouchardiere C, Desseigne F, Wang Q, Attignon V, Fondrevelle ME, De La Fouchardiere A, Perol M, Cassier P, Seigne C, Perol D, Ray-Coquard I, Meeus P, Fayette J, Flechon A, Le Cesne A, Penel N, Tredan O, Blay JY. The sum of gains and losses of genes encoding the protein tyrosine kinase targets predicts response to multi-kinase inhibitor treatment: Characterization, validation, and prognostic value. Oncotarget. 2015 Sep 22;6(28):26388-99. doi: 10.18632/oncotarget.4557. PMID 26317543